CLINICAL TRIAL: NCT05023434
Title: The Effect of Intraoperative Cortical Stimulation on Hand Strength and Function During Awake Craniotomies
Brief Title: A Study to Measure the Effect of Brain Stimulation on Hand Strength and Function in Patients With Brain Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Max Krucoff, MD, Assistant Professor of Neurological Surgery, Medical College of Wisconsin
Other Study IDs: PRO00040251
Record Dates: First submitted 2021-06-30; First posted 2021-08-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor; Brain Cancer; Motor Cortex; Lesion
Keywords: Brain Stimulation; Cortex Stimulation; Hand Motor Cortex; Primary Motor Cortex; M1; Resection; Surgery; Healthy Volunteers; Hand Strength; Hand Function
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Awake Craniotomy
  Interventions: Procedure: Intraoperative Brain Simulation - Alternate Stimulation Parameters
- Healthy Volunteers - No Longer Enrolling

INTERVENTIONS:
Procedure: Intraoperative Brain Simulation - Alternate Stimulation Parameters — Additional stimulation parameters outside of standard of care during intraoperative brain stimulation to aid in motor mapping.
  Groups: Awake Craniotomy

SUMMARY:
The neurosurgical standard of care for treating a patient with a tumor invading hand primary motor cortex (M1) includes performing a craniotomy with intraoperative direct electrical stimulation (DES) mapping and to resect as much tumor as possible without a resultant permanent neurological deficit. However, the subjective nature of current intraoperative hand motor assessments do not offer a comprehensive understanding of how hand strength and function may be impacted by resection. Additionally, there is a paucity of data to inform how altering DES parameters may effect motor mapping. Here, the investigators seek to demonstrate a feasible, standardized protocol to quantitatively assess hand strength and function and systematically assess several stimulation parameters to improve intraoperative measurements and better understand how cortical stimulation interacts with underlying neural function.

ELIGIBILITY:
AWAKE CRANIOTOMY COHORT

Inclusion Criteria:

1. Age 18 - 75
2. Ability to understand a written informed consent document, and the willingness to sign it
3. Radiographic evidence of tumor on MRI (i.e. non-enhancing) invading primary motor cortex in the non-dominant hemisphere.
4. Karnofsky performance status (KPS) ≥ 70
5. Normal or near normal motor strength (i.e., at least 3/5 in relevant areas)
6. Normal or near normal speech (Can consistently name at least 4/5 cards)
7. Free of other illness, in the judgment of the investigator, that may shorten life expectancy
8. Willing and able to participate in all aspects of the study

Exclusion Criteria:

1. Presence of other malignancy not in remission
2. Evidence of bi-hemispheric or widespread tumor involvement
3. Medically high-risk surgical candidate
4. History of recent scalp or systemic infection
5. Presence of other implants or foreign bodies in the head
6. Inability to receive an MRI for any reason
7. Inability to receive cortical stimulation for any reason
8. Presence of implanted cardiac device (such as a pacemaker or defibrillator)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a clinical indication for an awake craniotomy with motor mapping.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hand strength - Manual Motor Scale (0-5) | Pre-op, intra-op, 1 week post-op and 3 months post-op; 2 visits 3 weeks apart for healthy volunteers
  Quantitative assessment on a scale of 0 - 5 5 - normal strength 4 - give away weakness 3 - movement against gravity 2 - movement in anti-gravity position 1 - muscle twitch 0 - no movement
Change in Hand strength - Dynamometer grip and pinch strength (Newtons) | Pre-op, intra-op, 1 week post-op and 3 months post-op; 2 visits 3 weeks apart for healthy volunteers
  Scored using force production in kilograms (0-90) Standardized procedure for positioning
Chang in Hand function (Velocity) | Pre-op, intra-op, 1 week post-op and 3 months post-op; 2 visits 3 weeks apart for healthy volunteers
  The Cyberglove III collects data on the movement of the joints in the hand. Subjects will be asked to wear the Cyberglove III while doing various tasks. Velocity will be measured in degrees per second.
Chang in Hand function (Finger Individuation) | Pre-op, intra-op, 1 week post-op and 3 months post-op; 2 visits 3 weeks apart for healthy volunteers
  The Cyberglove III collects data on the movement of the joints in the hand. Subjects will be asked to wear the Cyberglove III while doing various tasks. Finger individuation will be calculated using joint angles.
Chang in Hand function (Smoothness) | Pre-op, intra-op, 1 week post-op and 3 months post-op; 2 visits 3 weeks apart for healthy volunteers
  The Cyberglove III collects data on the movement of the joints in the hand. Subjects will be asked to wear the Cyberglove III while doing various tasks. Smoothness will be calculated using joint angles.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No